CLINICAL TRIAL: NCT02875886
Title: DD-study: Diet or Diuretics for Salt-sensitivity in Chronic Kidney Disease
Acronym: DD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Ewout Hoorn, Internist nephrologist, Erasmus Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NL54748.078.15
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Amiloride; Hydrochlorothiazide; Diet, Sodium-Restricted

ARMS (2):
- Diuretic treatment (Active Comparator): Patients receive amiloride and hydrochlorothiazide
  Interventions: Drug: Amiloride; Drug: Hydrochlorothiazide
- Low-sodium diet (Active Comparator): Patients are put on a low-sodium diet (60 mmol/day)
  Interventions: Other: Low-sodium diet

INTERVENTIONS:
Drug: Amiloride — Combined with hydrochlorothiazide
  Arms: Diuretic treatment
Drug: Hydrochlorothiazide — Combined with amiloride
  Arms: Diuretic treatment
Other: Low-sodium diet
  Arms: Low-sodium diet

SUMMARY:
In this clinical study the anti-hypertensive response to dietary salt restriction is compared with the anti-hypertensive response to the diuretics hydrochlorothiazide/amiloride in adult patients with chronic kidney disease.

DETAILED DESCRIPTION:
Patients with chronic kidney disease (CKD) are exquisitely salt-sensitive. Salt-sensitivity in CKD is linked to hypertension and cardiovascular outcomes. Dietary salt restriction is an accepted intervention for salt-sensitivity in CKD. Another strategy, however, could be to block sodium uptake by the kidney pharmacologically by diuretics. Especially diuretics acting on the distal tubule may be effective, because this appears to be the site of increased sodium reabsorption in CKD. It is currently unknown how these two strategies, diet or diuretics, relate. The investigators hypothesize that diuretics are non-inferior to diet.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* CKD stage 3 or 4 (MDRD-GFR 15-60 ml/min)
* Use of any anti-hypertensive drugs
* No anti-hypertensive drugs but an average office systolic blood pressure > 140 mmHg (as measured by datascope)

Exclusion Criteria:

* Salt-wasting CKD
* Nephrotic syndrome
* Pregnant or breastfeeding women
* Life expectancy < 6 months
* Severe heart failure (NYHA III or IV) or liver cirrhosis with ascites and the inability to withdraw diuretics
* Rapidly declining kidney function with high likelihood of dialysis or kidney transplantation in the coming 4 months
* Kidney transplant recipients
* Use of immunosuppressive drugs
* Use of non-steroidal anti-inflammatory drugs
* Previous intolerance or allergy to hydrochlorothiazide or amiloride
* Serum sodium < 135 mmol/l
* Serum potassium < 3.5 mmol/l or > 5.0 mmol/l
* Inability to adhere to the study protocol (due to language, incapacitated subjects, subjects with intellectual disability)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-09; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
24 hour blood pressure | Two weeks after start of each intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ewout J Hoorn, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- ErasmusMC, Rotterdam, Netherlands

REFERENCES:
- [Background] Meng L, Fu B, Zhang T, Han Z, Yang M. Salt sensitivity of blood pressure in non-dialysis patients with chronic kidney disease. Ren Fail. 2014 Apr;36(3):345-50. doi: 10.3109/0886022X.2013.866008. Epub 2013 Dec 17. PMID 24345270
- [Background] McMahon EJ, Campbell KL, Bauer JD, Mudge DW. Altered dietary salt intake for people with chronic kidney disease. Cochrane Database Syst Rev. 2015 Feb 18;(2):CD010070. doi: 10.1002/14651858.CD010070.pub2. PMID 25691262
- [Background] Agarwal R, Sinha AD, Pappas MK, Ammous F. Chlorthalidone for poorly controlled hypertension in chronic kidney disease: an interventional pilot study. Am J Nephrol. 2014;39(2):171-82. doi: 10.1159/000358603. Epub 2014 Feb 11. PMID 24526255
- [Background] Slagman MC, Nguyen TQ, Waanders F, Vogt L, Hemmelder MH, Laverman GD, Goldschmeding R, Navis G. Effects of antiproteinuric intervention on elevated connective tissue growth factor (CTGF/CCN-2) plasma and urine levels in nondiabetic nephropathy. Clin J Am Soc Nephrol. 2011 Aug;6(8):1845-50. doi: 10.2215/CJN.08190910. Epub 2011 Jul 22. PMID 21784839
- [Background] Levy Yeyati N, Fellet A, Arranz C, Balaszczuk AM, Adrogue HJ. Amiloride-sensitive and amiloride-insensitive kaliuresis in advanced chronic kidney disease. J Nephrol. 2008 Jan-Feb;21(1):93-8. PMID 18264941
- [Derived] McMahon EJ, Campbell KL, Bauer JD, Mudge DW, Kelly JT. Altered dietary salt intake for people with chronic kidney disease. Cochrane Database Syst Rev. 2021 Jun 24;6(6):CD010070. doi: 10.1002/14651858.CD010070.pub3. PMID 34164803
- [Derived] Bovee DM, Visser WJ, Middel I, De Mik-van Egmond A, Greupink R, Masereeuw R, Russel FGM, Danser AHJ, Zietse R, Hoorn EJ. A Randomized Trial of Distal Diuretics versus Dietary Sodium Restriction for Hypertension in Chronic Kidney Disease. J Am Soc Nephrol. 2020 Mar;31(3):650-662. doi: 10.1681/ASN.2019090905. Epub 2020 Jan 29. PMID 31996411